CLINICAL TRIAL: NCT03693300
Title: A Phase II, Open-Label, Multi-Centre, International Safety Study of Durvalumab Following Sequential Chemotherapy and Radiation Therapy in Patients With Stage III, Unresectable Non-Small Cell Lung Cancer (PACIFIC 6)
Brief Title: A Study to Determine Safety of Durvalumab After Sequential Chemo Radiation in Patients With Unresectable Stage III Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4194C00006; 2018-002220-16 (EudraCT Number)
Record Dates: First submitted 2018-09-11; First posted 2018-10-02 (Actual); Results first posted 2022-10-07 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-05

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: Stage III Non-Small Cell Lung Cancer; Durvalumab; IV infusion immunoglobulin G (IgG); Antibody-dependent cellular cytotoxicity; Complement-dependent cytotoxicity; Monotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- WHO/ECOG PS 0 to 1 Cohort (Experimental): 100-120 participants will receive 1500 mg Durvalumab (MEDI4736) monotherapy via IV infusion q4w for up to a maximum of 24 months (up to 26 doses/cycles) with the last administration at Week 104. The study drug should be discontinued prior to 24 months if there is clinical progression or confirmed radiological progression or if there is unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met.
  Interventions: Drug: Durvalumab
- WHO/ECOG PS 2 Cohort (Experimental): up to 30 participants will receive 1500 mg Durvalumab (MEDI4736) monotherapy via IV infusion q4w for up to a maximum of 24 months (up to 26 doses/cycles) with the last administration at Week 104. The study drug should be discontinued prior to 24 months if there is clinical progression or confirmed radiological progression or if there is unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met.
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — Participants will receive 1500 mg Durvalumab monotherapy via IV infusion q4w for up to a maximum of 24 months with the last administration at Week 104.
  Other Names: MEDI4736

SUMMARY:
This is a Phase II, open-label, multi-centre study to determine the safety of a fixed dose of Durvalumab (MEDI4736) (1500 mg) every 4 weeks [q4w] in participants with unresectable Stage III Non-Small Cell Lung Cancer (NSCLC), who have not progressed following platinum-based sequential chemoradiation therapy (sCRT). This study will be conducted in Europe and North America.

DETAILED DESCRIPTION:
This is a Phase II, open-label, multi-centre study to determine safety of a fixed dose of Durvalumab (MEDI4736) (1500 mg) monotherapy in participants with unresectable Stage III NSCLC who have not progressed following definitive, platinum-based sCRT. Approximately, 150 participants will be treated with the study drug in Europe and North America. Participants will be in complete response (CR), partial response (PR), or have stable disease (SD) following definitive, platinum-based sCRT, as assessed by the Investigator and further supported by the screening imaging radiological assessment. Participants must not have progressed following definitive, platinum-based sCRT; radiation therapy must be completed within 42 days prior to first Investigational product (IP) dose administration. Participants must have histologically- or cytologically-documented NSCLC and locally-advanced, unresectable Stage III disease. Participants will be treated with the study drug in 2 cohorts: approximately 100-120 participants in the World Health Organization/Eastern Cooperative Oncology Group Performance Status (WHO/ECOG PS) 0 to 1 Cohort and up to 30 participants in the WHO/ECOG PS 2 Cohort.

ELIGIBILITY:
Inclusion criteria:

1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
2. Provision of signed and dated, written ICF prior to any mandatory study specific procedures, sampling, and analyses.
3. Provision of signed and dated written genetic informed consent prior to collection of sample for genetic analysis (optional).
4. 18 years or older at the time of signing the ICF.
5. Histologically- or cytologically-documented NSCLC with locally-advanced, unresectable Stage III disease (according to the IASLC Staging Manual Version 8 [IASLC 2016]). Positron emission tomography (PET)/CT, MRI of the brain, and endobronchial ultrasound with biopsy are highly encouraged at diagnosis.
6. Receipt of sCRT which must have been completed within 42 days prior to first IP dose administration in the study.

   1. The platinum-based chemotherapy regimen must contain cisplatin or carboplatin and 1 of the following agents: etoposide, vinblastine, vinorelbine, a taxane (paclitaxel or docetaxel), or pemetrexed, according to the local standard of care (SoC) regimens. Platinum-based chemotherapy containing cisplatin or carboplatin and gemcitabine is permitted under certain conditions - refer to bullet point 6(b).
   2. Patients must have received at least 2 cycles of platinum-based chemotherapy before radiation therapy. The interval between administration of the last dose of chemotherapy regimen and start of radiation therapy must be no more than 6 weeks. Consolidation chemotherapy after radiation is not permitted.

   (i) If the patient's platinum-based chemotherapy contained gemcitabine, no overlap between chemotherapy and radiation therapy is permitted.

   (ii) If the patient's platinum-based chemotherapy contained any of the agents listed in (a) other than gemcitabine, an overlap of 1 cycle of chemotherapy and radiation therapy is acceptable.

   (c) Patients must have received a total dose of radiation of 60 Gy ±10% (54 Gy to 66 Gy). Sites are encouraged to adhere to mean organ radiation dosing as follows: (i) Mean lung dose <20 Gy and/or V20 <35%; (ii) Mean oesophagus <34 Gy; (iii) Heart V45 <35% or V30 <30%. Note: Sites should be aware of the recent RTOG 0617 Study data demonstrating that doses higher than 60 Gy may be associated with greater toxicity and worse efficacy.

   (d) Patients with WHO/ECOG PS 2 or chronic lung disease (pulmonary emphysema or chronic obstructive pulmonary disease) must have received a V20 <25%.
7. Patients must not have progressed following platinum-based sCRT, as per Investigator assessed RECIST 1.1 criteria. . In order to assess disease progression, the baseline imaging (CT/MRI) used for Screening purposes should be compared against the most recently performed scan that allows physician assessment as per RECIST 1.1 criteria. If an intermediate scan taken between chemotherapy and radiotherapy is available and that scan is suitable for physician assessment as per RECIST 1.1 criteria, then this scan should be used.

   1. Patients with measurable disease and/or non-measurable and/or no evidence of disease (NED) assessed at baseline by CT/MRI will be entered in this study.
   2. Prior irradiated lesions may be considered measurable and selected as TLs provided they fulfil the other criteria for measurability.
8. Must have a life expectancy of at least 12 weeks at enrolment.
9. WHO/ECOG PS ≤2.
10. Adequate organ and marrow function at enrolment as defined below. These parameters should be achieved without augmentation by growth factors, transfusions, or infusions within 14 days of screening unless required for SoC:

    1. Haemoglobin ≥9.0 g/dL;
    2. Absolute neutrophil count >1.0 × 109/L;
    3. Platelet count >75 × 109/L;
    4. Serum bilirubin ≤1.5 × upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome, who will be allowed in consultation with their physician.
    5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN.
    6. Measured creatinine clearance >40 mL/min or calculated creatinine clearance >40 mL/min as determined by Cockcroft-Gault (using actual body weight) (Cockcroft and Gault 1976).

Males:

Creatinine clearance (mL/min) = Weight (kg) × (140 Age) 72 × serum creatinine (mg/dL)

Females:

Creatinine clearance (mL/min) = Weight (kg) × (140 Age) × 0.85 72 × serum creatinine (mg/dL)

11 Body weight >30 kg at enrolment and first IP dose administration. 12 Male or female. 13 Evidence of post-menopausal status, or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

1. Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
2. Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).

Exclusion criteria:

1. Patients with locally-advanced NSCLC whose disease has progressed following platinum based sCRT.
2. Patients who have disease considered for surgical treatment as part of their care plan, such as Pancoast or superior sulcus tumours.
3. Mixed small-cell lung cancer and NSCLC histology.
4. History of allogeneic organ transplantation.
5. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

   1. Patients with vitiligo or alopecia.
   2. Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement.
   3. Any chronic skin condition that does not require systemic therapy.
   4. Patients without active disease in the last 5 years at enrolment may be included but only after consultation with the Study Physician.
   5. Patients with celiac disease controlled by diet alone.
6. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, ILD, serious chronic GI conditions associated with diarrhoea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs, or compromise the ability of the patient to give written informed consent.
7. History of another primary malignancy except for:

   1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence.
   2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
   3. Adequately treated carcinoma in situ without evidence of disease.
8. History of leptomeningeal carcinomatosis.
9. History of active primary immunodeficiency.
10. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), hepatitis B (known positive hepatitis B surface antigen [HbsAg] result), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies). Patients with a past or resolved hepatitis B virus (HBV) infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HbsAg) are eligible. Patients positive for hepatitis C antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA).
11. Any unresolved toxicity of NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.

    1. Patients with Grade ≥2 neuropathy or Grade ≥2 lymphopenia will be evaluated on a case-by-case basis after consultation with the Study Physician.
    2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab (MEDI4736) may be included only after consultation with the Study Physician.
12. Known allergy or hypersensitivity to durvalumab (MEDI4736) or any of the IP excipients.
13. Patients who have received cCRT for locally-advanced NSCLC, or who received sCRT with at least 2 concomitant CRT cycles. Prior surgical resection (ie, Stage I or II) is permitted.

    Note: Patients whose platinum-based chemotherapy contained gemcitabine and who received sCRT with at least 1 concomitant CRT cycle are excluded from this study.
14. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP.

    Note: Patients, if enrolled, should not receive live vaccine while receiving IP and up to 30 days after the last dose of IP.
15. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP.

    Note: Local surgery of isolated lesions for palliative intent is acceptable.
16. Prior exposure to immune-mediated therapy, including but not limited to, other anti CTLA-4, anti-PD-1, anti-PD-L1, and anti PD L2 antibodies, excluding therapeutic anticancer vaccines.
17. Current or prior use of immunosuppressive medication within 14 days before the first dose of IP. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra articular injection);
    2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent;
    3. Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication).
18. Previous IP assignment in the present study.
19. Concurrent enrolment in another clinical study, unless it is an observational (noninterventional) clinical study or the follow-up period of an interventional study.
20. Participation in another clinical study with an IP during the 4 weeks prior to the first IP dose administration.
21. Prior randomisation or treatment in a previous durvalumab (MEDI4736) ± tremelimumab clinical study regardless of treatment arm assignment.
22. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of IP.
23. Judgment by the Investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions, and requirements.
24. Genetic research study (optional):

Exclusion criteria for participation in the optional (DNA) genetic research component of the study include:

1. Previous allogeneic bone marrow transplant.
2. Non-leukocyte-depleted whole blood transfusion in 120 days of genetic sample collection.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2023-04-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (2):
  - Research Site, Gainesville, Georgia
  - Research Site, Knoxville, Tennessee
- France (4):
  - Research Site, Créteil
  - Research Site, Paris
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Toulouse
- Germany (5):
  - Research Site, Gauting
  - Research Site, Großhansdorf
  - Research Site, Hamm
  - Research Site, Hanover
  - Research Site, Heidelberg
- Italy (6):
  - Research Site, Avellino
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Monza
  - Research Site, Parma
  - Research Site, Roma
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Guadalajara
  - Research Site, Madrid
  - Research Site, Seville
  - Research Site, Valencia
- United Kingdom (6):
  - Research Site, Leeds
  - Research Site, Manchester
  - Research Site, Middlesbrough
  - Research Site, Nottingham
  - Research Site, Sheffield
  - Research Site, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Garassino MC, Mazieres J, Reck M, Chouaid C, Bischoff H, Reinmuth N, Cove-Smith L, Mansy T, Cortinovis D, Migliorino MR, Delmonte A, Sanchez JG, Chara Velarde LE, Bernabe R, Paz-Ares L, Perez ID, Trunova N, Foroutanpour K, Faivre-Finn C. Durvalumab After Sequential Chemoradiotherapy in Stage III, Unresectable NSCLC: The Phase 2 PACIFIC-6 Trial. J Thorac Oncol. 2022 Dec;17(12):1415-1427. doi: 10.1016/j.jtho.2022.07.1148. Epub 2022 Aug 9. PMID 35961520
- See also: CSP Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4194C00006&attachmentIdentifier=223d186d-4d3f-48ae-992c-86d35a9632c5&fileName=AZ_D4194C00006-csp-v4_Redacted_PDF_A.pdf&versionIdentifier=
- See also: SAP Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4194C00006&attachmentIdentifier=03fb15bd-8baa-46db-808c-d332d239328f&fileName=AZ_D4194C00006-sap-ed-5__Redacted_PDF_A.pdf&versionIdentifier=
- See also: CSR Synopsis Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4194C00006&attachmentIdentifier=829673e0-d101-44cf-81e3-fb3a2f283905&fileName=AZ_D4194C00006-study-synopsis_Redacted_PDF_A.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 16 April 2019 to 21 April 2023 at 25 sites in the United States of America (USA), France, Germany, Italy, Spain, and the United Kingdom.
Pre-assignment Details: Patients who met all the inclusion and none of the exclusion criteria were included in the study. The screening period was from Day -28 to Day -1. The Study was scheduled from initiation of durvalumab up to a maximum of 24 months of treatment, 3 months of safety follow up and subsequent survival follow up as per CSP. Informed consent form was signed prior to screening procedures.
Groups:
- Durvalumab Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1: Patients received 1500 mg Durvalumab monotherapy via Intravenous (IV) infusion every 4 weeks (q4w).
- Durvalumab ECOG PS 2: Patients received 1500 mg Durvalumab monotherapy via IV infusion q4w.
Period: Overall Study
Arm/Group | Durvalumab Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1 | Durvalumab ECOG PS 2
Started | 114 | 3
Completed | 56 | 1
Not Completed | 58 | 2
Not completed — Withdrawal by Subject | 6 | 0
Not completed — Death | 50 | 2
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set consisted of all patients who received at least one dose of (partial or in full) of study drug.
Groups:
- Durvalumab ECOG PS 0 or 1; Durvalumab ECOG PS 2: Patients received 1500 mg Durvalumab monotherapy via IV infusion q4w.
- Total: Total of all reporting groups
Arm/Group | Durvalumab ECOG PS 0 or 1 | Durvalumab ECOG PS 2 | Total
Number analyzed (Participants) | 114 | 3 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (8.46) | 65.0 (12.00) | 66.9 (8.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 1 | 44
  Male | 71 | 2 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 103 | 3 | 106
  Unknown or Not Reported | 10 | 0 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 101 | 3 | 104
  Unknown | 13 | 0 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Grade 3 and Grade 4 Treatment-related Adverse Events (TRAEs)
Description: Safety and tolerability of Durvalumab as defined by Grade 3 and Grade 4 TRAEs following IV infusion administration was assessed.
Time Frame: Up to 6 months
Population: The safety analysis set consisted of all patients who received at least one dose of IP (partial or in full).
Measure: Count of Participants; unit: Participants
Groups:
- Durvalumab Total: Patients received 1500 mg Durvalumab monotherapy via IV infusion q4w.
Arm/Group | Durvalumab ECOG PS 0 or 1 | Durvalumab ECOG PS 2 | Durvalumab Total
Number analyzed (Participants) | 114 | 3 | 117
Participants
  Any possibly related AEs of CTCAE Grade 3 or Grade 4 | 7 | 0 | 7
  Any possibly related AEs of Grade 3 or Grade 4 with onset date within 6 months of the first dose | 5 | 0 | 5
Statistical Analysis 1: Comparison: Durvalumab ECOG PS 0 or 1; Any possibly related adverse events of CTCAE Grade 3 or Grade 4; Test type: Other; Proportion (%) = 6.1, 95% CI 2-sided [2.50 to 12.24] — 95% CI were based on the Clopper-Pearson method
Statistical Analysis 2: Comparison: Durvalumab ECOG PS 2; Any possibly related adverse events of CTCAE Grade 3 or Grade 4; Test type: Other; Proportion (%) = 0, 95% CI 2-sided [0.00 to 70.76] — 95% CI were based on the Clopper-Pearson method
Statistical Analysis 3: Comparison: Durvalumab Total; Any possibly related adverse events of CTCAE Grade 3 or Grade 4; Test type: Other; Proportion (%) = 6.0, 95% CI 2-sided [2.44 to 11.94] — 95% CI were based on the Clopper-Pearson method
Statistical Analysis 4: Comparison: Durvalumab ECOG PS 0 or 1; Any possibly related AEs of Grade 3 or Grade 4 with onset date within 6 months of the first dose; Test type: Other; Proportion (%) = 4.4, 95% CI 2-sided [1.44 to 9.94] — 95% CI were based on the Clopper-Pearson method
Statistical Analysis 5: Comparison: Durvalumab ECOG PS 2; Any possibly related AEs of Grade 3 or Grade 4 with onset date within 6 months of the first dose; Test type: Other; Proportion (%) = 0, 95% CI 2-sided [0.00 to 70.76] — 95% CI were based on the Clopper-Pearson method
Statistical Analysis 6: Comparison: Durvalumab Total; Any possibly related AEs of Grade 3 or Grade 4 with onset date within 6 months of the first dose; Test type: Other; Proportion (%) = 4.3, 95% CI 2-sided [1.40 to 9.69] — 95% CI were based on the Clopper-Pearson method

2. Secondary Outcome: Progression-free Survival (PFS)
Description: The efficacy of Durvalumab (MEDI4736) treatment in terms of PFS. PFS was defined as the time from the first date of treatment until the date of objective disease progression based on Investigator's assessment according to RECIST 1.1 or death (by any cause in the absence of progression) regardless of whether the patient withdraws from IP or receives another anticancer therapy prior to progression.
Time Frame: From the first date of treatment until the date of objective disease progression or death (approximately upto 48 months)
Population: The safety analysis set consisted of all patients who received at least one dose of IP (partial or in full).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab ECOG PS 0 or 1 | Durvalumab ECOG PS 2 | Durvalumab Total
Number analyzed (Participants) | 114 | 3 | 117
Months | 13.1 [7.36 to 19.91] | 3.7 [1.81 to NA] — Not calculated due to low number of events as well as low sample size. | 13.1 [7.36 to 19.91]

3. Secondary Outcome: Percentage of Patients Progression-free at 12 Months
Description: The percentage of patients treated with Durvalumab who are progression-free was estimated. PFS12 according to RECIST 1.1 as assessed by the Investigator.
Time Frame: From the first date of treatment until the date of objective disease progression or death (upto 12 months)
Population: The safety analysis set consisted of all patients who received at least one dose of IP (partial or in full).
Measure: Number (95% Confidence Interval); unit: Percentage of patient
Arm/Group | Durvalumab ECOG PS 0 or 1 | Durvalumab ECOG PS 2 | Durvalumab Total
Number analyzed (Participants) | 114 | 3 | 117
Percentage of patient | 51.1 [41.29 to 60.02] | 33.3 [0.90 to 77.41] | 50.6 [40.97 to 59.45]

4. Secondary Outcome: Overall Survival (OS)
Description: The efficacy of Durvalumab (MEDI4736) treatment in terms of OS were assessed. OS was defined as the time from the first date of treatment until death due to any cause. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive.
Time Frame: From the first date of treatment until death due to any cause (approximately upto 48 months)
Population: The safety analysis set consisted of all patients who received at least one dose of IP (partial or in full).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab ECOG PS 0 or 1 | Durvalumab ECOG PS 2 | Durvalumab Total
Number analyzed (Participants) | 114 | 3 | 117
Months | 39.0 [30.59 to NA] — Not calculated due to insufficient number of events. | 12.3 [4.96 to NA] — Not calculated due to insufficient number of events. | 39.0 [30.59 to NA] — Not calculated due to insufficient number of events.

5. Secondary Outcome: Percentage of Patients Alive
Description: Percentage of patients alive at 12 months, 24 months, and 36 months were estimated.
Time Frame: From the first date of treatment until the date of objective disease progression or death (12 months, 24 months, and 36 months)
Population: The safety analysis set consisted of all patients who received at least one dose of IP (partial or in full).
Measure: Number (95% Confidence Interval); unit: Percentage of patient
Arm/Group | Durvalumab ECOG PS 0 or 1 | Durvalumab ECOG PS 2 | Durvalumab Total
Number analyzed (Participants) | 114 | 3 | 117
Percentage of patient
  Survival at 12 months | 83.9 [75.73 to 89.57] | 66.7 [5.41 to 94.52] | 83.5 [75.36 to 89.15]
  Survival at 24 months | 68.2 [58.54 to 76.00] | 33.3 [0.90 to 77.41] | 67.2 [57.73 to 75.08]
  Survival at 36 months | 57.2 [46.94 to 66.20] | NA [NA to NA] — Not calculated due to insufficient number of events. | 56.5 [46.41 to 65.46]

6. Secondary Outcome: Objective Response Rate (ORR)
Description: The efficacy of Durvalumab (MEDI4736) treatment in terms of ORR were assessed. ORR (based on Investigator assessed response to treatment of complete response (CR) and partial response (PR) as per RECIST 1.1 criteria), together with the corresponding 95% CI, was reported for patients. Objective response is complete response (CR), or partial response (PR) confirmed by a follow-up visit at least 4 weeks after. Both visits contributing to response should have occurred before any further anti-cancer therapy, in order for the patient to be considered a responder. Responses that occurred after the start of subsequent anti-cancer therapy were not included in the numerator. Response excluded unconfirmed response. Participants with unconfirmed responses include those whose CR, or PR don't have a confirmed response. These responses occur at any time during the study, recur after anti-cancer therapy, and these participants were missing for a follow-up visit 4 weeks after.
Time Frame: From 8 weeks ±1 week after investigational product (IP) treatment initiation and continue every 8 weeks (q8w) ±1 week through 52 weeks and every 12 weeks (q12w) ±1 week until disease progression (approximately upto 48 months)
Population: The safety analysis set consisted of all patients who received at least one dose of IP (partial or in full). Patients without a post-baseline assessment were not included.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab ECOG PS 0 or 1 | Durvalumab ECOG PS 2 | Durvalumab Total
Number analyzed (Participants) | 114 | 3 | 117
Participants
  Number of patients with response | 24 | 0 | 24
  Number of patients with unconfirmed response | 5 | 0 | 5

7. Secondary Outcome: Duration of Response (DOR) From Onset of Response
Description: The efficacy of Durvalumab (MEDI4736) treatment in terms of DoR were assessed. DoR was defined as the time from the date of first documented response per RECIST1.1 until the first date of documented progression per RECIST1.1 or death in the absence of disease progression. If a patient did not progress following a response, then the patients' DoR was censored at the PFS censoring time.
Time Frame: From 8 weeks ±1 week after IP treatment initiation and continue q8w ±1 week through 52 weeks and q12w ±1 week until disease progression (approximately upto 48 months)
Population: The safety analysis set consisted of all patients who received at least one dose of IP (partial or in full). The patients with objective response were evaluated.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Durvalumab ECOG PS 0 or 1 | Durvalumab ECOG PS 2 | Durvalumab Total
Number analyzed (Participants) | 24 | 0 | 24
Weeks | NA [NA to NA] — Not calculated due to insufficient number of events. |  | NA [NA to NA] — Not calculated due to insufficient number of events.

8. Secondary Outcome: Lung Cancer Mortality
Description: The efficacy of durvalumab (MEDI4736) treatment in terms of lung cancer mortality was assessed. Lung Cancer Mortality was defined as the time from the date of treatment start until death due to lung cancer. Any patient not known to have died due to lung cancer will be censored based on the last recorded date on which the patient was known to be alive or died due to reason other than lung cancer.
Time Frame: From date of treatment start until death due to lung cancer (approximately upto 48 months)
Population: The safety analysis set consisted of all patients who received at least one dose of IP (partial or in full). Patients who had died due to causes related to non-small cell lung cancer were evaluated.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab ECOG PS 0 or 1 | Durvalumab ECOG PS 2 | Durvalumab Total
Number analyzed (Participants) | 40 | 1 | 41
Months | 41.8 [36.50 to NA] — Not calculated due to insufficient number of events. | NA [4.96 to NA] — Not calculated due to insufficient number of events. | 41.8 [36.50 to NA] — Not calculated due to insufficient number of events.

9. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Event of Special Interests (AESIs), and Immune-mediated Adverse Event (imAEs)
Description: The safety and tolerability profile of Durvalumab(MEDI4736) treatment, including all AEs were assessed.
Time Frame: Until the final visit (upto 48 months)
Population: The safety analysis set consisted of all patients who received at least one dose of IP (partial or in full). This include treatment emergent AEs only, ie. AEs occurred during screening period are NOT included.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab ECOG PS 0 or 1 | Durvalumab ECOG PS 2 | Durvalumab Total
Number analyzed (Participants) | 114 | 3 | 117
Participants
  Any AE | 108 | 3 | 111
  Any AE possibly related to treatment | 87 | 3 | 90
  Any AE of CTCAE Grade 3 or Grade 4 | 32 | 0 | 32
  Any AE of CTCAE Grade 3 or Grade 4, possibly related to treatment | 7 | 0 | 7
  Any AE with outcome of death | 3 | 0 | 3
  Any AE with outcome of death, possibly related to treatment | 1 | 0 | 1
  Any SAE (including events with outcome of death) | 32 | 0 | 32
  Any SAE (including events with outcome of death), possibly related to treatment | 7 | 0 | 7
  Any AE leading to discontinuation of treatment | 32 | 0 | 32
  Any AE leading to discontinuation of treatment, possibly related to treatment | 19 | 0 | 19
  Any AE leading to treatment interruption | 52 | 1 | 53
  Any AE leading to treatment interruption, possibly related to treatment | 24 | 1 | 25
  Any AESI or AEPI (including events with outcome of death) | 86 | 3 | 89
  Any AESI or AEPI (including events with outcome of death), possibly related to treatment | 73 | 2 | 75
  Any imAE | 48 | 2 | 50
  Any imAE, possibly related to treatment | 43 | 2 | 45
  Any imAE as assessed by Investigator | 64 | 1 | 65
  Any imAE as assessed by Investigator, possibly related to treatment | 64 | 1 | 65

ADVERSE EVENTS:
Time Frame: Upto 48 months
Arm/Group | Durvalumab ECOG PS 0 or 1 | Durvalumab ECOG PS 2 | Durvalumab Total
All-Cause Mortality (participants affected / at risk) | 50/114 | 2/3 | 52/117
Serious Adverse Events (participants affected / at risk) | 32/114 | 0/3 | 32/117
Other Adverse Events (participants affected / at risk) | 106/114 | 3/3 | 109/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab ECOG PS 0 or 1 (N=114) | Durvalumab ECOG PS 2 (N=3) | Durvalumab Total (N=117)
Pneumonia (Infections and infestations) | 5 (7) | 0 (0) | 5 (7)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (2) | 0 (0) | 1 (2)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 5 (5)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 1 (3)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (2) | 0 (0) | 1 (2)
Cardiac failure (Cardiac disorders) | 1 (2) | 0 (0) | 1 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab ECOG PS 0 or 1 (N=114) | Durvalumab ECOG PS 2 (N=3) | Durvalumab Total (N=117)
Pneumonia (Infections and infestations) | 8 (8) | 0 (0) | 8 (8)
Nasopharyngitis (Infections and infestations) | 10 (12) | 0 (0) | 10 (12)
Hypothyroidism (Endocrine disorders) | 15 (15) | 1 (1) | 16 (16)
Hyperthyroidism (Endocrine disorders) | 12 (12) | 0 (0) | 12 (12)
Decreased appetite (Metabolism and nutrition disorders) | 14 (14) | 1 (2) | 15 (16)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (8) | 1 (1) | 8 (9)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (6) | 0 (0) | 6 (6)
Insomnia (Psychiatric disorders) | 7 (7) | 0 (0) | 7 (7)
Headache (Nervous system disorders) | 17 (18) | 1 (1) | 18 (19)
Paraesthesia (Nervous system disorders) | 9 (9) | 0 (0) | 9 (9)
Hypertension (Vascular disorders) | 7 (8) | 1 (2) | 8 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 43 (49) | 2 (3) | 45 (52)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 (39) | 2 (3) | 29 (42)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 16 (20) | 1 (1) | 17 (21)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 0 (0) | 10 (11)
Constipation (Gastrointestinal disorders) | 23 (24) | 0 (0) | 23 (24)
Diarrhoea (Gastrointestinal disorders) | 24 (33) | 0 (0) | 24 (33)
Nausea (Gastrointestinal disorders) | 17 (21) | 0 (0) | 17 (21)
Vomiting (Gastrointestinal disorders) | 9 (9) | 0 (0) | 9 (9)
Dry mouth (Gastrointestinal disorders) | 7 (7) | 0 (0) | 7 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 19 (21) | 2 (3) | 21 (24)
Rash (Skin and subcutaneous tissue disorders) | 13 (17) | 1 (1) | 14 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 (28) | 1 (2) | 23 (30)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (17) | 0 (0) | 17 (17)
Asthenia (General disorders) | 29 (40) | 2 (2) | 31 (42)
Fatigue (General disorders) | 24 (35) | 0 (0) | 24 (35)
Pyrexia (General disorders) | 22 (25) | 0 (0) | 22 (25)
Non-cardiac chest pain (General disorders) | 15 (18) | 1 (1) | 16 (19)
Oedema peripheral (General disorders) | 10 (10) | 0 (0) | 10 (10)
Blood creatinine increased (Investigations) | 8 (13) | 0 (0) | 8 (13)
Gamma-glutamyltransferase increased (Investigations) | 7 (9) | 0 (0) | 7 (9)
Alanine aminotransferase increased (Investigations) | 6 (7) | 0 (0) | 6 (7)
Weight decreased (Investigations) | 8 (8) | 0 (0) | 8 (8)
Conjunctivitis (Infections and infestations) | 4 (4) | 0 (0) | 4 (4)
Lower respiratory tract infection (Infections and infestations) | 4 (6) | 0 (0) | 4 (6)
Oral candidiasis (Infections and infestations) | 4 (4) | 0 (0) | 4 (4)
Urinary tract infection (Infections and infestations) | 5 (5) | 0 (0) | 5 (5)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 6 (6) | 0 (0) | 6 (6)
Depressed mood (Psychiatric disorders) | 4 (4) | 0 (0) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 6 (8) | 0 (0) | 6 (8)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 6 (8) | 0 (0) | 6 (8)
Vertigo (Ear and labyrinth disorders) | 4 (5) | 0 (0) | 4 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 0 (0) | 6 (8)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 0 (0) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 6 (6) | 0 (0) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 0 (0) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (5) | 0 (0) | 5 (5)
Noninfective gingivitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 4 (4)
Erythema (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 4 (4)
Night sweats (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 4 (4)
Psoriasis (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0) | 4 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0) | 4 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 3 (4)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 3 (3) | 0 (0) | 3 (3)
Chills (General disorders) | 3 (3) | 0 (0) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 3 (3) | 0 (0) | 3 (3)
Blood thyroid stimulating hormone increased (Investigations) | 4 (4) | 0 (0) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 3 (4)
COVID-19 (Infections and infestations) | 7 (7) | 0 (0) | 7 (7)
Rhinitis (Infections and infestations) | 3 (3) | 0 (0) | 3 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 3 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (6) | 0 (0) | 3 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 4 (4)
Depression (Psychiatric disorders) | 3 (3) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 7 (13) | 0 (0) | 7 (13)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 3 (3) | 0 (0) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 3 (3)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 4 (4)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 3 (4) | 0 (0) | 3 (4)
Rash pruritic (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 3 (3)
Chest pain (General disorders) | 3 (3) | 0 (0) | 3 (3)
Blood glucose increased (Investigations) | 3 (3) | 0 (0) | 3 (3)
Lipase increased (Investigations) | 3 (4) | 0 (0) | 3 (4)
Platelet count decreased (Investigations) | 3 (4) | 0 (0) | 3 (4)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document contains trade secrets and confidential commercial information, disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (2):
  • Study Protocol (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT03693300/Prot_002.pdf
  • Statistical Analysis Plan (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT03693300/SAP_003.pdf